CLINICAL TRIAL: NCT05575583
Title: Clinical Study of Repeated Transcranial Magnetic Stimulation in the Prevention and Treatment of Postoperative Executive Dysfunction
Brief Title: rTMS in the Prevention and Treatment of Postoperative Executive Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuzhou Central Hospital (Other)
Collaborators: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: XuzhouCH20221001
Record Dates: First submitted 2022-09-29; First posted 2022-10-12 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2022-09

CONDITIONS: Executive Function Disorder; Functional Magnetic Resonance Imaging
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Subjects underwent repetitive transcranial magnetic stimulation for five consecutive days from day 2 to day 6 after surgery. The stimulation target area was the posterior cingulate gyrus, and the neuronavigation system was used to accurately locate the stimulation target in this project. Continuous theta short rapid pulse mode (cTBS) was used. CTBS mode consisted of a slave stimulus delivered every 0.2 seconds (5Hz), and each slave stimulus consisted of three bursts of 50Hz. A single stimulus lasts about 40 seconds and totals 600 pulses. Stimulation sessions are from 8 to 10 a.m. daily.
  Interventions: Device: repetitive transcranial magnetic stimulation
- Control group (Sham Comparator): Subjects underwent repetitive transcranial magnetic stimulation for five consecutive days from day 2 to day 6 after surgery，but the machine does not turn on.
  Interventions: Device: pseudo repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — The neural navigation system was used to accurately locate the stimulus target.Continuous theta short rapid pulse mode was used. CTBS mode consisted of a slave stimulus delivered every 0.2 seconds (5Hz), and each slave stimulus consisted of three bursts of 50Hz. A single stimulus lasts about 40 seconds and totals 600 pulses.
  Arms: Intervention group
Device: pseudo repetitive transcranial magnetic stimulation — Participant in control group receive pseudo repetitive transcranial magnetic stimulation
  Arms: Control group

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) is a new neuroelectrophysiological technique developed in recent years. rTMS can affect local and distant cortical function, promote regional reconstruction of cortical function, and has clear curative effect on a variety of neuropsychiatric diseases. Previous study found that rTMS can improve postoperative cognitive function, and there may be a dual biological mechanism. Brain network abnormalities may be the direct cause of postoperative cognitive dysfunction, and neuroinflammation is one of the key molecular mechanisms behind postoperative cognitive dysfunction . rTMS may play a role in the regulation of brain network and inflammatory molecules, and thus play a role in the prevention and treatment of postoperative cognitive dysfunction (POCD).

DETAILED DESCRIPTION:
This study intends to use neuroimaging methods to observe the correlation between neuroinflammation and brain network abnormalities in patients with POCD, and verify the repair effect of rTMS intervention on the pathological changes, so as to provide a theoretical basis for further optimizing the establishment of rTMS localization therapy model for POCD.

ELIGIBILITY:
Inclusion Criteria:

* Heart valve replacement.
* 45 to 75 years old.

Exclusion Criteria:

* definite cerebral infarction.
* failure and decompensation of vital organs
* physical metal implants.
* severe neuropsychiatric disorders.
* less than 9 years of education.
* alcohol abuse.
* drug dependence.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Stroop color words test(SCWT) | Preoperative
  The Stroop Color Words test (SCWT) was used to evaluate the dominant inhibition in executive function
Trail making test | Preoperative
  Trail Making test (TMT) was used to evaluate the set switching in executive function
Corsi Block test | Preoperative
  The visuospatial working memory of executive function was assessed by the Corsi Block test
Stroop color words test(SCWT) | Postoperative 1 week
  The Stroop Color Words test (SCWT) was used to evaluate the dominant inhibition in executive function
Trail making test | Postoperative 1 week
  Trail Making test (TMT) was used to evaluate the set switching in executive function
Corsi Block test | Postoperative 1 week
  The visuospatial working memory of executive function was assessed by the Corsi Block test

SECONDARY OUTCOMES:
Functional magnetic resonance brain network characteristics | Preoperative
  The changes of brain network between intervention group and control group before and after operation were compared. Resting-state fMRI and task-state fMRI were evaluated.
Functional magnetic resonance brain network characteristics | Postoperative 1 week
  The changes of brain network between intervention group and control group before and after operation were compared. Resting-state fMRI and task-state fMRI were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Yangzi Zhu, Doctor, Principal Investigator — Xuzhou Central Hospital; Liwei Wang, Doctor, Study Director — Xuzhou Central Hospital; Qi Yang, Doctor, Study Director — Beijing Chao Yang Hospital; Daqing Ma, Study Chair — Imperial College London, Chelsea and Westminster Hospital
Locations (1):
- Xuzhou Central Hospital, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No